CLINICAL TRIAL: NCT00443508
Title: Reduction or Discontinuation of Calcineurine Inhibitors With Conversion to Everolimus-Based Immunosuppresion to Alleviate Chronic Allograft Nephropathy (CAN) in Kidney Transplant Recipients: A Prospective Randomized Study
Brief Title: Reduction or Discontinuation of CNI's With Conversion to Everolimus-Based Immunosuppresion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001AIL01
Record Dates: First submitted 2007-03-04; First posted 2007-03-06 (Estimated); Last update posted 2007-03-06 (Estimated); Status verified 2005-09

CONDITIONS: Kidney Diseases
Keywords: everolimus; renal transplant; tacrolimus; Certican; CHRONIC ALLOGRAFT NEPHROPATHY; Renal transplant patients
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: adding Certican to therapy
Drug: reducing Tacrolimus

SUMMARY:
This study is design to compare two different strategies aiming to lessen the degree of the ongoing process of allograft injury either by removing tacrolimus from the maintenance immunosuppressive protocol or by reducing tacrolimus dose.

The primary goal is to assess the change in renal function at 6 and 12 months after conversion using creatinine levels and calculated creatinine clearance.

The study will include two groups: The study group of 30 patients and a matched control group with creatinine levels at similar range.

DETAILED DESCRIPTION:
This study is design to compare two different strategies aiming to lessen the degree of the ongoing process of allograft injury either by removing tacrolimus from the maintenance immunosuppressive protocol or by reducing tacrolimus dose.

The primary goal is to assess the change in renal function at 6 and 12 months after conversion using creatinine levels and calculated creatinine clearance.

The study will include two groups: The study group of 30 patients and a matched control group with creatinine levels at similar range.

Patients will undergo the following baseline studies:

1. Doppler ultrasound to exclude any mechanical or a vascular problem.
2. A kidney biopsy to define the histological changes (degree of interstitial fibrosis, tubular and glomerular changes). The biopsies will be stained also for C4D and for fibrinogenic markers (TGF-beta, and collagen).
3. A 24-hour urine protein excretion and creatinine clearance
4. Echocardiography study
5. Carotid Ultrasound

The following parameters will be monitored every clinic visit throughout the study period:

1. SMA-12 including creatinine levels.
2. A complete blood count.
3. Cholesterol, HDL-cholesterol and triglyceride levels.
4. Blood pressure measurements (X2)
5. The number of blood pressure medications.
6. Cholesterol lowering medication requirement
7. Urine protein excretion (quantitative spot-test )
8. Protein amount in the urine

Study end points:

The data will be evaluated based on an intention to treat analysis and the following parameters will be compared between the two groups:

1. Creatinine levels and calculated creatinine clearance
2. Spot urine for Cr./protein ratio
3. 24-hr. protein excretion
4. Change in peak diastolic and mean arterial blood pressure
5. The number and dosage of blood pressure medications
6. Cholesterol, HDL and triglyceride levels
7. Proportion of patients on cholesterol lowering agents
8. Number and severity of biopsy proven acute rejection episodes
9. Incidence of biopsy proven chronic rejection. (depends on per protocol biopsy at end of study)
10. Patient and graft survival

ELIGIBILITY:
Inclusion Criteria:

* Patients on CNI FK < 5 ng/m"l with MPA / Imuran with or without steroids
* Renal impairment GFR between 30 - 70 m"l/minute/
* Patient who signed Informed consent
* Patient with no contraindication to renal biopsy
* Women who are not pregnant and will use contraception

Exclusion Criteria:

* Proteinuria > 100 m"g/mmol Creatinine
* Acute rejection during 3 months before screening
* WBC < 2500, plt < 50,000,
* Nephropathy due to polyoma virus
* Patients on other investigational drugs
* Patients on rapamycin
* Patients with HIV or other systemic infection
* Inability to comply with protocol requirements
* Active or history of malignancy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2007-02; Study Completion 2010-02

PRIMARY OUTCOMES:
The primary goal is to assess the change in renal function
at 6 and 12 months after conversion using creatinine levels
and calculated creatinine clearance.

SECONDARY OUTCOMES:
The secondary aim is to assess changes in cardiovascular risks at
12 months after conversion (glucose control., cholesterol and
triglyceride levels and hypertension control), incidence of
acute and chronic rejection and graft and patient survival rates.

CONTACTS AND LOCATIONS:
Overall Officials: Eytan Mor, Prof, Principal Investigator — Rabin Medical Center, head of Transplantation department
Locations (1):
- Transplantation department, rabin Medical Center, Petah Tikva, Israel